CLINICAL TRIAL: NCT01405677
Title: A Phase II Open, Randomised, Controlled Study to Evaluate the Safety and Immunogenicity of a Paediatric Dose (0.25 mL) and the Standard Dose (0.5 mL) of Epaxal® With Reference to Havrix Junior® Healthy in Healthy Children and Adolescents (>=12 Months - 16 Years of Age) Using a 0/6 Month Schedule
Brief Title: Safety and Immunogenicity of a Paediatric Dose of Virosomal Hepatitis A Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EPA 001 FU
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2013-12

CONDITIONS: Hepatitis A
Keywords: Hepatitis A; Vaccination; Immunisation
MeSH Terms: conditions — Hepatitis A | interventions — epaxal berna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Epaxal 0.25 mL (Experimental): Single intramuscular dose (M. deltoideus) given on Day 1 and at Month 6
  Interventions: Biological: Epaxal 0.25 mL
- Epaxal 0.5 mL (Active Comparator): Single intramuscular dose (M. deltoideus) given on Day 1 and at Month 6
  Interventions: Biological: Epaxal 0.5 mL
- Havrix Junior (Active Comparator): Single intramuscular dose (M. deltoideus) given on Day 1 and at Month 6
  Interventions: Biological: Havrix Junior 0.5 mL

INTERVENTIONS:
Biological: Epaxal 0.25 mL — 12 IU hepatitis A antigen coupled to immunopotentiating reconstituted Influenza virosome (IRIV)
  Arms: Epaxal 0.25 mL
Biological: Epaxal 0.5 mL — 24 IU hepatitis A antigen coupled to IRIV
  Arms: Epaxal 0.5 mL
Biological: Havrix Junior 0.5 mL — 720 EU hepatitis A antigen absorbed onto aluminum hydroxide
  Arms: Havrix Junior

SUMMARY:
The primary purpose of the original study was to assess whether the protection afforded by the paediatric dose of Epaxal vaccine against hepatitis A was not inferior to the protection afforded by the standard dose of Epaxal. The aim of the follow-up phase was to perform a computer based modelling analysis of the long term protection afforded by the paediatric dose, and to compare this with the standard dose and also with an alternative hepatitis A vaccine (Havrix Junior).

ELIGIBILITY:
Inclusion Criteria:

Original study:

* Males or females aged >=12 months and 16 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject when applicable and from the parent/legal guardian of the subject. - Free of obvious health problems as established by medical history and/or clinical examination before entering the study.

Follow up phase:

* Subjects enrolled and randomized in the primary study and having received two doses of the study vaccine

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period and safety follow-up
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. (For corticosteroids, this means prednisone, or equivalent, >=0.5 mg/kg/day. Inhaled and topical steroids were allowed.)
* Planned administration/administration of a vaccine not foreseen by the study protocol within 4 weeks prior to the first dose of study vaccine
* Previous vaccination against hepatitis A
* Seropositive for anti-HAV antibodies (>=10 mIU/mL)
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness
* Acute disease at the time of enrolment

Ages: 12 Months to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 308 (Actual)
Dates: Start 2004-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Individual anti-HAV titers | 66 months post-booster
  Real-time seroprotection analysis and computer modelling will be conducted up to 5 years post-booster to estimate long term seroprotection
Individual anti-HAV titers | 18 months post-booster
  Real-time seroprotection analysis and computer modelling will be conducted up to 5 years post-booster to estimate long term seroprotection
Individual anti-HAV titers | 30 months post-booster
  Real-time seroprotection analysis and computer modelling will be conducted up to 5 years post-booster to estimate long term seroprotection
Individual anti-HAV titers | 42 months post-booster
  Real-time seroprotection analysis and computer modelling will be conducted up to 5 years post-booster to estimate long term seroprotection
Individual anti-HAV titers | 54 months post-booster
  Real-time seroprotection analysis and computer modelling will be conducted up to 5 years post-booster to estimate long term seroprotection

SECONDARY OUTCOMES:
Geometric mean titers | 18, 30, 42, 54, 66 months post-booster
Seroprotection | 18, 30, 42, 54, 66 months post-booster
  Porportion of subjects who are seroprotected calculated at each time point where seroprotection is defined as >=10 mIU/mL

CONTACTS AND LOCATIONS:
Overall Officials: Pierre van Damme, MD, Principal Investigator — Universiteit Antwerpen; Andre Vertruyen, MD, Principal Investigator — Sint-Vincentiusziekenhuis
Locations (2):
- Belgium (2):
  - Sint-Vincentiusziekenhuis, Antwerp
  - Centre for the Evaluation of Vaccination, University of Antwerp, Antwerp